CLINICAL TRIAL: NCT06852365
Title: Resistant Starch Usage in Polycystic Ovary Syndrome: Impact on Cardiometabolic Dysfunction and the Gut Microbiome (CORS-PCOS)
Brief Title: Combined Oral Contraceptive Pill and Resistance Starch
Acronym: COR-PCOS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Anuja Dokras, Founder's Professor in Women's Health, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 856886; 1R01HL173772-01 (NIH)
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Metabolic Syndrome; Polycystic Ovary Syndrome
MeSH Terms: conditions — Metabolic Syndrome; Polycystic Ovary Syndrome | interventions — Contraceptives, Oral; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resistant Starch (Active Comparator): wheat dextrin
  Interventions: Dietary Supplement: wheat dextrin; Drug: Oral Contraceptives, Low-Dose
- Placebo (Placebo Comparator): maltodextrin
  Interventions: Drug: Oral Contraceptives, Low-Dose; Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: wheat dextrin — participants will take 15 grams per day for 12 weeks
  Other Names: Benefiber
  Arms: Resistant Starch
Drug: Oral Contraceptives, Low-Dose — 20 micrograms ethinyl estradiol and desogestrel 0.15mg
Dietary Supplement: Maltodextrin — participants will take 15 grams per day for 12 weeks
  Arms: Placebo

SUMMARY:
This study will enroll women with PCOS to study the effects of first line therapy, oral contraceptive pills, and then either 12 weeks of resistant starch or 12 weeks of placebo to explore if resistant starch improves cardiometabolic parameters or impacts gut dysbiosis compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Women between ages of 18-40 years with BMI greater than or equal to 25 kg/m² to less than or equal to 48 kg/m² diagnosed with PCOS defined by the Rotterdam criteria based on a history of chronic anovulation (8 or fewer periods), androgen excess [defined as total serum testosterone, free testosterone or a FAI greater than or equal to 90% of the upper limit of normal) or hirsutism (Ferriman-Gallwey score greater than 6 for Hispanics/ Black and greater than or equal to 2 for women of Asian descent)] and polycystic ovaries as defined by a pelvic ultrasound (20 or more follicles or ovarian vol greater than 10cm3) or elevated AMH.
2. For women with more regular bleeding patterns, but who are suspected to be experiencing periodic anovulatory bleeding, a midluteal progesterone (P4) level less than 3ng/dL will be evidence of ovulatory dysfunction and qualify as anovulation.
3. Women with only hyperandrogenic PCOS phenotype (hyperandrogenism + one more criteria) will be included to decrease the heterogeneity of the cohort and as metabolic risks are increased in these women compared to normo-androgenic women with PCOS.
4. Subjects should be willing to avoid pregnancy for the entire duration of the study.

Exclusion Criteria:

1. Subjects with other causes for irregular menses such as pregnancy, lactation, untreated hypothyroidism, untreated hyperprolactinemia and premature menopause.
2. Subjects with late onset adrenal hyperplasia
3. Subjects with history of bariatric surgery
4. Those who are unable to comply with the study procedures, for instance due to mental illness, substance abuse, or participation in other studies.
5. Subjects taking medications that affect weight or metabolic parameters (e.g. lipid lowering medications).
6. History of Crohn's disease and ulcerative colitis as well as current use of probiotics and laxatives are excluded.
7. Subjects could not have taken antibiotics for at least 3 months prior to randomization visit.
8. Subjects with greater than 20 g/day of dietary fiber intake based on pre-screening ASA-24 survey will be excluded.
9. Subjects with medical conditions that are contraindications to use of OCP and other medical conditions such as:

   1. Type 1 or 2 diabetes
   2. liver disease or dysfunctional liver (AST/ALT greater than 2x normal or a total bilirubin greater than 2.5 mg/dL)
   3. renal disease (BUN greater than 30 mg/dL or serum creatinine greater than 1.4 mg/dL)
   4. severe anemia (hemoglobin less than 10 mg/dL)
   5. alcohol abuse
   6. poorly controlled hypertension
   7. TG greater than 250 mg/dl
   8. chronic inflammatory conditions such as psoriasis
   9. history of deep venous thrombosis, pulmonary embolus, or cerebrovascular accident; known heart disease (New York Heart Association Class II or higher)
   10. history of cervical carcinoma, endometrial carcinoma, or breast carcinoma, adrenal or ovarian tumor secreting androgens, and Cushing's syndrome -

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Change in LDL-C measure | Baseline and 12 weeks
Change in fasting glucose measure | Baseline and 12 weeks
Change in systolic blood pressure | Baseline and 12 weeks
Change in diastolic blood pressure | Baseline and 12 weeks
Change in BMI | Baseline and 12 weeks
Change in Bifidobacteria abundance measured by quantitative polymerase chain reaction (q-PCR) | Baseline and 12 weeks
Change in Single Chain Fatty Acids (SCFA) | Baseline and 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided